CLINICAL TRIAL: NCT03096353
Title: Sensory and Opioid Mechanisms of Affective Touch
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 170075; 17-AT-0075
Record Dates: First submitted 2017-03-29; First posted 2017-03-30 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-06

CONDITIONS: Pain; Touch
Keywords: NALOXONE; fMRI; Functional Magnetic Resonance Imaging (fMRI)
MeSH Terms: conditions — Pain | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Naloxone, then Placebo (Experimental): Day one - During MRI session participant underwent sensory stimulus testing followed by bolus and infusion doses of naloxone (0.05 mg/kg bodyweight). When infusion levels reached stability, sensory testing was performed again.
  Day two - During MRI session participant underwent sensory stimulus testing followed by bolus and infusion doses of normal saline. When infusion levels reached stability, sensory testing was performed again.
  Interventions: Other: Placebo; Drug: Naloxone
- Placebo, then Naloxone (Experimental): Day one - During MRI session participant underwent sensory stimulus testing followed by bolus and infusion doses of normal saline. When infusion levels reached stability, sensory testing was performed again.
  Day two - During MRI session participant underwent sensory stimulus testing followed by bolus and infusion doses of naloxone (0.05 mg/kg bodyweight). When infusion levels reached stability, sensory testing was performed again.
  Interventions: Other: Placebo; Drug: Naloxone

INTERVENTIONS:
Other: Placebo — saline
Drug: Naloxone — We will be using naloxone at normal clinical doses as the study drug. Naloxone is an opiate antagonist and has been used since the 1960 s to reverse the effects of opiate overdoses.

SUMMARY:
Background:

Medicines called opioids are used to treat pain. The body also produces opioids. These are called endorphins. Researchers want to learn more about how these natural opioids work. This might lead to new therapies for conditions like depression, anxiety, and chronic pain.

Objective:

To determine how opioids affect how pleasant or unpleasant it feels when the skin is touched, compressed, or heated.

Eligibility:

Healthy right-handed adults ages 18-50.

Design:

Participants will be screened under another protocol.

Participants will have 2 study visits with the same procedures, at least 1 day apart. Each visit will last 3-4 hours.

Participants will wear shorts or change into scrubs so researchers can test on their legs.

Participants will answer questions and have urine tests.

Participants will have a brain magnetic resonance imaging (MRI) scan. The scanner is a metal cylinder in a strong magnetic field. Participants will lie on a table that slides in and out of the cylinder. A device called a coil will be placed over the head.

During MRI, participants will have sensory testing. They will get several types of touch to the calf of the leg. These include gentle brushing of the skin, gentle compression of the calf with an inflation sleeve, and heat stimuli.

Participants will have an intravenous line placed each day. They will get naloxone 1 day and saline the other day. Participants will not be told which they get. Naloxone is a drug that blocks opioid receptors.

The MRI and sensory testing will then be repeated.

After each stimuli block, participants will rate the sensations as well as their mood and calmness/anxiety.

DETAILED DESCRIPTION:
Objective: Our recent pilot study found evidence suggesting that blocking endogenous opioid release increases the pleasantness associated with having the skin stroked. Deep pressure touch (observed in hugs and massage) also typically conveys a sense of pleasantness. This increased pleasantness contrasts with evidence that blocking endogenous opioid release increases pain. The current study will examine the role of endogenous opioids in the pleasantness of light skin stroking and deep pressure touch, and contrast it with their role in the unpleasantness of a painful heat stimulus. Further, it will examine the neural basis of observed perceptual changes, using fMRI. This study constitutes the first study of the K99 phase of a K99/R00 grant application recently submitted to National Center for Complementary and Integrative Health (NCCIH) by Dr. Laura Case.

Study Population: 30 healthy participants will be enrolled in the study.

Design: Participants will receive intravenous saline or intravenous naloxone on separate days to investigate the effect of mu-opioid antagonism on the intensity and pleasantness of superficial and deep affective touch and the intensity and unpleasantness of cutaneous heat pain. Using a double-blind cross-over design, functional Magnetic Resonance Imaging (fMRI) will be conducted during sensory testing before and after the infusion of each drug to examine the neural mediation of opioid effects on touch perception. Ratings of mood, anxiety, pain intensity, pleasantness/unpleasantness, wanting and liking will also be collected throughout the study session.

Outcome measures: We will compare subjective ratings (mood, calmness, anxiety, pleasantness, wanting, liking, pain intensity and unpleasantness) during naloxone and saline to: 1) Determine whether naloxone increases the pleasantness and/or intensity of affective touch (light brush and deep compression); 2) Determine whether naloxone increases the unpleasantness and/or intensity of cutaneous heat pain; 3) Determine the role of mood or anxiety changes in mediating the effect of endogenous opioids on these perceptual measures; 3) Determine changes in the brain activation related to these effects.

ELIGIBILITY:
-INCLUSION CRITERIA:

All subjects must be:

* Between 18 and 50 years old.
* Right-handed (on Edinburgh Handedness Inventory).
* Fluent in English.
* Able to provide written informed consent.

EXCLUSION CRITERIA:

Overall exclusion criteria for the study:

* Unable to comply with study procedures (or does not rate stimuli as tolerable) or unable to schedule visits promptly (including inability to schedule the second session within approximately 14 days of the first session)
* Pregnancy or breastfeeding.
* Use of recreational drugs in the past month (e.g., marijuana, methylenedioxymethamphetamine (MDMA, 'ecstasy' or 'Molly'), Lysergic acid diethylamide (LSD), cocaine, methamphetamine, heroin, prescription and/or opioids).
* Congenital lower limb deficiency or amputation.
* Peripheral neuropathy, dermatological condition such as scars or burns, or has had a tattoo in the testing region within the previous four weeks that might influence cutaneous sensibility.
* Women who consume more than 7 alcoholic beverages per week, and men who consume more than 14 drinks per week.
* Current chronic pain condition or has had chronic pain in the past year (painful condition lasting more than six months), including ongoing treatment with medications for neuropathic pain (e.g. gabapentin, tricyclic antidepressants, pregabalin, tramadol)
* Major medical condition, such as kidney, liver, cardiovascular (including blood clots, hypertension, preexisting cardiac arrhythmia), autonomic, pulmonary, or neurological problems (e.g., seizure disorder ) or a chronic systemic disease (e.g., diabetes).
* Current diagnosis or pharmacological treatment of psychiatric disorders such as major depression, major anxiety-related problems, post-traumatic stress syndrome, bipolar disorder, psychosis, attention-deficit/hyperactivity disorder or current or lifetime alcohol or substance abuse disorders (as identified in study #16-AT-0077)
* Participant has metal in his/her body which would make having an MRI scan unsafe, such as pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal workers may have.
* Participant is uncomfortable in small closed spaces (has claustrophobia) so that he/she would feel uncomfortable in the MRI machine or cannot lie comfortably flat on his/her back for up to 75 minutes in the MRI scanner.
* Participants weighs more than 550 lbs.
* Participant has taken any pain medication other than an over-the-counter NSAIDs or acetaminophen within the last month or for more than one month on a continual basis within last six months.
* Previous participation in 13-AT-0143 (related study).
* NIH employees who are subordinates, relatives, or co-workers of the investigators, or NCCIH Division of Intramural Research (DIR) employees.
* Participants using medications that play into opioid pathways (e.g. loperamide or dextromethorphan), that could potentially interact with naloxone (naltrexone, methylnaltrexone, droperidol, fenfluramine and clonidine)
* Participant using any herbal supplements (such as yohimbine) due to risk of unknown dangerous interaction as there is no data for herbal preparations and naloxone.
* Participant has allergies to naloxone or similar drugs.

EXCLUSION CRITERIA FOR INIDIVIDUAL STUDY SESSION:

* Has consumed alcohol within 24 hours, shows signs of alcohol withdrawal syndrome, or has behavioral signs of intoxication will be excluded immediately and not have the possibility to reschedule their session.
* Used topical pain-relieving creams in the testing area (e.g. methylsalicylate, capsaicin) within 24 hours of testing or used non-steroidal anti-inflammatory drugs (NSAIDS, e.g. aspirin, ibuprofen), acetaminophen, or naproxen within 3 days of testing*.

  * To be determined during the pre-session screening. Participants who cannot refrain from these activities may have their session rescheduled up to two times. If the participant is found non-compliant during the second rescheduled appointment, he or she will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bushnell, Ph.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-AT-0075.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 subject consented; one subject consented but did not start either arm of the study
Period: Period 1
Arm/Group | Naloxone, Then Placebo | Placebo, Then Naloxone
Started | 15 | 13
Completed | 12 | 12
Not Completed | 3 | 1
Period: Period 2
Arm/Group | Naloxone, Then Placebo | Placebo, Then Naloxone
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naloxone, Then Placebo | Placebo, Then Naloxone | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 4 | 9
  White | 4 | 6 | 10
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pleasantness of Skin Brushing From Before to After Infusion
Description: Measurement of brushing pleasantness using a visual analogue scale. Sensory hedonics (unpleasantness vs. pleasantness) was assessed on a scale ranging from extremely unpleasant (-100) to neutral (0), to extremely pleasant (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Naloxone: During MRI session participant underwent sensory stimulus testing followed by bolus and infusion doses of naloxone (0.05 mg/kg bodyweight). When infusion levels reached stability, sensory testing was performed again.
- Placebo: During MRI session participant underwent sensory stimulus testing followed by bolus and infusion doses of normal saline. When infusion levels reached stability, sensory testing was performed again.
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | -9.6875 (21.6314) | -4.9583 (22.3983)

2. Secondary Outcome: Changes in Pleasantness of Deep Skin Pressure From Before to After Infusion
Description: Measurement of pressure pleasantness/unpleasantness using a visual analogue scale. Sensory hedonics (unpleasantness vs. pleasantness) was assessed on a scale ranging from extremely unpleasant (-100) to neutral (0), to extremely pleasant (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | -2.25 (22.3527) | -1.375 (15.4196)

3. Secondary Outcome: Change in Unpleasantness of Cutaneous Heat Pain From Before to After Infusion
Description: Measurement of heat pleasantness/unpleasantness using a visual analogue scale. Sensory hedonics (unpleasantness vs. pleasantness) was assessed on a scale ranging from extremely unpleasant (-100) to neutral (0), to extremely pleasant (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | -5.75 (27.2969) | -3.4783 (26.2728)

4. Secondary Outcome: Changes in Intensity of Skin Brushing From Before to After Infusion
Description: Measurement of brushing intensity using a visual analogue scale. Intensity was assessed on a scale ranging from no sensation (-100) to pain threshold (0), to intolerable pain (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | -4.5833 (12.7511) | 4.7917 (23.3065)

5. Secondary Outcome: Changes in Intensity of Deep Skin Pressure From Before to After Infusion
Description: Measurement of pressure intensity using a visual analogue scale. Intensity was assessed on a scale ranging from no sensation (-100) to pain threshold (0), to intolerable pain (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | -3.8333 (21.2671) | -4 (20.4762)

6. Secondary Outcome: Changes in Intensity of Cutaneous Heat Pain From Before to After Infusion
Description: Measurement of heat intensity using a visual analogue scale. Intensity was assessed on a scale ranging from no sensation (-100) to pain threshold (0), to intolerable pain (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | 4.4583 (22.1970) | -1.3043 (24.6092)

7. Other Pre Specified Outcome: Activation in Somatosensory Cortex (S2) Brain Area of Interest (ROI) During Brushing
Description: Functional MRI Blood-oxygen-level-dependent (BOLD) activation in secondary somatosensory cortex (S2) during brushing. BOLD signal is typically expressed as arbitrary units (AU's) measured from "0 to 100% change". 0 being no change and 100% maximum change
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Arbitrary units | 0.0475 (32.5047) | 9.6547 (31.2841)

8. Other Pre Specified Outcome: Activation in Somatosensory Cortex (S2) Brain Area of Interest (ROI) During Pressure
Description: Functional MRI Blood-oxygen-level-dependent (BOLD) activation in secondary somatosensory cortex (S2) during pressure. BOLD signal is typically expressed as arbitrary units (AU's) measured from "0 to 100% change". 0 being no change and 100% maximum change
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Arbitrary units | -3.1585 (42.3639) | 17.4139 (32.5070)

9. Other Pre Specified Outcome: Changes in Mood During Skin Brushing From Before to After Infusion
Description: Mood during brushing was assessed using a visual analogue scale ranging from extremely bad mood (-100) to neutral mood (0), to extremely good mood (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | -2.375 (19.0652) | 1.16667 (17.5537)

10. Other Pre Specified Outcome: Changes in Mood During Skin Pressure From Before to After Infusion
Description: Mood during skin pressure was assessed using a visual analogue scale ranging from extremely bad mood (-100) to neutral mood (0), to extremely good mood (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | 3.2083 (20.8287) | -1.7917 (28.6657)

11. Other Pre Specified Outcome: Changes in Mood During Cutaneous Heat From Before to After Infusion
Description: Mood during heat was assessed using a visual analogue scale ranging from extremely bad mood (-100) to neutral mood (0), to extremely good mood (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | 0.3333 (21.0717) | -5.3478 (20.7476)

12. Other Pre Specified Outcome: Changes in Anxiety During Skin Brushing From Before to After Infusion
Description: Anxiety during brushing was assessed using a visual analog scale ranging from extreme anxiety (-100) to neutral (0) to extreme calm (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | -2.7917 (21.8197) | -8.5 (22.4304)

13. Other Pre Specified Outcome: Changes in Anxiety During Deep Skin Pressure From Before to After Infusion
Description: Anxiety during pressure was assessed using a visual analog scale ranging from extreme anxiety (-100) to neutral (0) to extreme calm (100).
Time Frame: One day, within a 2 hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | 0.0417 (28.3568) | -5.9167 (12.7392)

14. Other Pre Specified Outcome: Changes in Anxiety During Cutaneous Heat From Before to After Infusion
Description: Anxiety during heat was assessed using a visual analog scale ranging from extreme anxiety (-100) to neutral (0) to extreme calm (100).
Time Frame: One day, within a 2-hour session
Population: All participants who completed both the treatment and placebo phases of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 24 | 24
Units on a scale | 4.0833 (22.2583) | -12.0435 (19.3654)

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Naloxone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT03096353/Prot_SAP_000.pdf